CLINICAL TRIAL: NCT02502058
Title: Observational, Case-Series Study Evaluation of Bone Width and Dental Implant Stability When Using the Densah Bur™ Bone Compaction Process to Prepare Dental Implant Sites
Brief Title: Dental Implant Stability When Using the Densah Bur™ Bone Compaction Process to Prepare Dental Implant Sites
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left her employment at the University.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: University_of_Minnesota2
Record Dates: First submitted 2015-07-10; First posted 2015-07-17 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Densah Bur™ , osseodensification — Densah™ bur (Versah Osseodensification Company™) is used to prepare dental implant sites, in human subjects, by compacting (osseodensification ) bone vs. removing bone to create the opening in the jaw bone into which the dental implant is then placed. This osseodensification process results in increased bone-ridge width, increased compact bone in the outer wall of the prepared sites, and; it is believed, increases implant stability.
  Other Names: Versah Osseodensification Company™

SUMMARY:
The primary objective of this study is to determine if the use of a bone compaction process (osseodensification) (Densah™ bur: Versah Osseodensification Company™) to prepare dental implant sites, in human subjects, results in increased bone-ridge width, increased compact bone in the outer wall of the prepared sites, and dental implant stability.

DETAILED DESCRIPTION:
The proposed project will be an observational, case-series study. The investigators anticipate enrolling 40 study subjects. Treatment Procedures: Following initial treatment planning discussions between the dentists and their patients regarding all of their dental treatment options, those patients who opt to have dental implants placed will be approached to discuss participation in the current study. Before entry into the study, the Investigator or an authorized member of the investigational staff will explain to potential subjects the aims, methods, reasonable anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the subject will receive for the treatment of their condition. Subjects will be told that alternative treatments are available and that if they decline to take part in the present study that such a refusal will not prejudice future treatment. Those patients who are willing to participate will be scheduled for their initial and follow-up dental implant visits at the School of Dentistry. At the baseline visit the study outcome data will be collected; including: 1) measuring the bone-ridge width, before and after implant site preparation (drilling); 2) intraoral photographs of the prepared opening; 3) dental implant torque readings will be obtained; and 4) ISQ as measure of both initial and the dynamic development of osseointegration (the formation of a direct interface between the dental implant and bone) over time. The ISQ measurements will be collected again at three and six-weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Ages 18-80 years of age
3. Missing at least one tooth.
4. Capable of giving informed consent

Exclusion Criteria:

1. Patient is a pregnant female
2. Patient smoking more than 5 cigarettes per day
3. Patient has a history of alcoholism or drug abuse during the last 5 years
4. Patient with uncontrolled hypertension or diabetes
5. Patient has a malignant tumor
6. Patient is on daily dose of steroids
7. Patient with history of chemotherapy or radiation for the last 12 months
8. Patient who is immuno suppressed
9. Patient with titanium allergy
10. Subject should not be a homeless person

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study subjects will include 40 healthy adult patients who seek dental implant placement to replace missing teeth in their mouths.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Bone-ridge width before and immediately after preparation of the implant site when using the Densah Bur. | intraoperative
  The width of the bony ridge into which the dental implant will be placed will be measured immediately before drilling the opening with the Densah Bur and then again following completion of drilling but before the dental implant is placed into the prepared opening. These measurements will occur at the time of the implant surgery.

SECONDARY OUTCOMES:
insertion torque value (ITV) | intraoperative
  ITV is a measure of the rotational friction between the implant and the surrounding bone
implant stability quotient (ISQ) | intraoperative , at 3 weeks and 6 weeks post surgery
  ISQ uses resonance frequency analysis to determine if the newly prepared implant site is stable enough for immediate or early loading of the actual dental implant.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Lenton, MA, Principal Investigator — University of Minnesota
Locations (1):
- Oral Health Research Clinic at the School of Dentistry at the University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share study data.

REFERENCES:
- See also: Website for the manufacturer of the Densah Bur Technology — http://versah.com